CLINICAL TRIAL: NCT03074539
Title: Sleep-Disordered Breathing in Chronic Thromboembolic Pulmonary Hypertension - a Prospective, Descriptive Cohort Study
Brief Title: Sleep-Disordered Breathing in Chronic Thromboembolic Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Klaus Hackner, MD, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTEPH_SDB
Record Dates: First submitted 2017-02-14; First posted 2017-03-08 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulmonary Endarteriectomy - PEA (Active Comparator): CTEPH treatment via PEA. This arm includes patients who will receive Pulmonary Endarteriectomy (PEA) according to local CTEPH board recommendation. A standardized polygraphy will be conducted before the PEA - intervention, to obtain information concerning Sleep Disorder Breathing. 6 months after the PEA surgery another polygraphy will be accomplished and the results compared with the first polygraphy and the other arms.
  If Sleep Disorder Breathing remains, a personalized recommendation on further specific therapy (e.g. nocturnal continuous positive airway pressure ventilation) will be made.
  Interventions: Procedure: Pulmonary Endarteriectomy
- Balloon Pulmonary Angioplasty - BPA (Active Comparator): CTEPH treatment via BPA. Patients who are suitable for Balloon Pulmonary Angioplasty (BPA) according to the recommendation of the local CTEPH board (e.g. patients not suitable for Pulmonary Endarteriectomy). A standardized polygraphy will be conducted before the first BPA intervention, to gain information about possible sleep-disordered breathing. 6 months after the first BPA intervention another polygraphy will be accomplished and the results compared with the first polygraphy and the other arms.
  If Sleep Disorder Breathing remains, a personalized recommendation on further specific therapy (e.g. nocturnal continuous positive airway pressure ventilation) will be made.
  Interventions: Procedure: Ballon Pulmonary Angioplasty
- Medical Treatment (Active Comparator): CTEPH treatment via Medical Treatment. Patients who are inoperable (not suitable for Pulmonary Endarteriectomy) and not eligible for BPA according to the recommendation of the local CTEPH board will get medical treatment with Riociguat. The treatment will be assigned according to the currently valid guidelines (2015 European Respiratory Society / European Society of Cardiology guidelines on the diagnosis and treatment of pulmonary hypertension). A standardized polygraphy will be conducted before the medical treatment starts, another polygraphy will be conducted after 6 months of treatment if Riociguat. The results will be compared with the first polygraphy and the other arms.
  If Sleep Disorder Breathing remains, a personalized recommendation on further specific therapy (e.g. nocturnal continuous positive airway pressure ventilation) will be made.
  Interventions: Drug: Riociguat

INTERVENTIONS:
Drug: Riociguat — Patients will be treated with Riociguat according to guidelines (2015 ERS/ESC guidelines for the diagnosis and treatment of pulmonary hypertension) and manufacturers recommendation.
  Other Names: Adempas
  Arms: Medical Treatment
Procedure: Pulmonary Endarteriectomy — Patients will receive Pulmonary Endarteriectomy if they are suitable for this procedure according to the recommendation of the local CTEPH board. Patients must also consent to this surgical procedure.
  Other Names: PEA
  Arms: Pulmonary Endarteriectomy - PEA
Procedure: Ballon Pulmonary Angioplasty — Patients will receive Ballon Pulmonary Angioplasty if they are suitable for this procedure according to the recommendation of the local CTEPH board (e.g. not suitable for PEA). Patients must also consent to this procedure.The BPA will be accomplished in several interventions.
  Other Names: BPA
  Arms: Balloon Pulmonary Angioplasty - BPA

SUMMARY:
There is evidence for a high prevalence of Sleep Disorder Breathing (SDB) in patients with Chronic Thromboembolic Pulmonary Hypertension (CTEPH). Central Sleep Apnea, Cheyne-Stokes Breathing and Obstructive Sleep Apnea appear to occur in CTEPH. However, there is no information on the impact of CTEPH treatment modalities on concomitant SDB. Furthermore, the use of PAP therapy in CTEPH has not yet been investigated. CTEPH is a rare and serious disease and there may be a bidirectional association of SDB and CTEPH.

This study plans to investigate the prevalence of SDB in CTEPH and compare it to datasets of large epidemiological studies on SDB. Furthermore, the impact of CTEPH treatment on SDB will be analyzed and CTEPH patients for possible PAP treatment will be defined.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed untreated CTEPH
* NYHA I-III

Exclusion Criteria:

* Age<18
* Pulmonary Hypertension other than CTEPH
* Previous diagnosis of SDB
* Ongoing PAP treatment
* Use of nasal oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
AHI change under CTEPH treatment | 6 months
  Change from baseline AHI (Apnoe-Hypopnoe Index, events/h) after 6 months of CTEPH treatment

SECONDARY OUTCOMES:
Number of patients with persisting elevated AHI (= ≥15/h) after CTEPH treatment | Time point: 6 months after the individual start of the CTEPH treatment
  Patients with persisting elevated AHI will be assessed for further PAP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Irene Lang, Prof., Study Chair — Medical University Vienna
Locations (1):
- Medical Unviersity Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided